CLINICAL TRIAL: NCT00134940
Title: A Non-interventional Protocol to Collect Prospective and Retrospective Data in Patients Receiving Everolimus to Prevent Acute Rejection Following Cardiac Transplantation
Brief Title: Post-marketing Study to Collect Safety Data in Heart Transplant Patients Receiving Everolimus
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Other Study IDs: CRAD001A2424
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Heart Disease
Keywords: Transplantation, heart; Organ transplant
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort

SUMMARY:
The purpose of this observational protocol is to evaluate the use of everolimus in routine clinical practice for heart transplants.

Primary outcome measures: incidence of acute rejection episodes Secondary outcomes: safety

ELIGIBILITY:
Inclusion Criteria:

* Cardiac transplant recipients
* Discharged alive from hospital
* Must be receiving everolimus

Exclusion Criteria:

* Patients not treated with everolimus beginning within 2 weeks after receiving a heart transplant

Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (6):
- Austria (3):
  - Novarits, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis, Wein
- Germany (3):
  - Novartis, Bad Oeynhausen
  - Novartis Investigative Site, Berlin
  - Novartis, Erlangen